CLINICAL TRIAL: NCT01291316
Title: GABAergic Modulation in Pain Transmission in Human: Effect of the GABAA Agonist Clobazam on Peripheral and Central Sensitisation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jules Desmeules, MD, University Hospital, Geneva
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GABA-SPUM
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Clonazepam; Tolterodine Tartrate; Clobazam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- clobazam (Experimental)
  Interventions: Drug: clobazam
- clonazepam (Active Comparator)
  Interventions: Drug: Clonazepam
- tolterodine (Placebo Comparator)
  Interventions: Drug: Tolterodine

INTERVENTIONS:
Drug: Clonazepam — clonazepam, 1 mg, single oral dose
  Arms: clonazepam
Drug: Tolterodine — Tolterodine 1,37mg, single oral dose
  Arms: tolterodine
Drug: clobazam — clobazam 20 mg, single oral dose
  Arms: clobazam

SUMMARY:
In animal, the GABAergic system modulates central sensitisation, which is a key phenomenon in pain processing. The development of GABAA agonists targeting the subunits of the GABAA receptor implicated in nociception, but not the subunit implicated in sedation is attractive as it opens new perspectives of testing the role of GABAergic modulation of pain processing in human volunteers. The purpose of this subproject is to test the effect of the specific α2 and α3 agonist but sparing α1 effect TPA023 on a human model of peripheral and central sensitisation and to correlate its pharmacodynamic effect with the pharmacokinetic of the compound.

The results would contribute to clarify the potential role of these α2/α3 agonist but sparing α1drugs in clinical pain conditions.

DETAILED DESCRIPTION:
Objectives:

* To assess the effect of the GABAA agonist clobazam on central sensitisation (change in the size of the area of secondary hyperalgesia) in healthy volunteers.
* To assess the effect of the GABAA agonist clobazam on peripheral sensitisation.
* To assess the effect of the GABAA agonist clobazam on sedation.
* To correlate the pharmacokinetic of clobazam to its effect (PK-PD modelling)
* To describe the role of the polymorphisms of CYP450 2C19 in the pharmacokinetic and dynamic of clobazam.

Methodology :

phase II , exploratory, three arms randomised placebo-controlled, double blind cross-over study in healthy volunteers

Number of patients : 25

Test product,Dose, Route of administration :

Clobazam,20 mg,oral intake

Duration of treatment :

Single dose administration of each compound

Reference therapy :

Clonazepam 1mg, oral intake Tolterodine 1, 37mg, oral intake

Other therapy :

Flumazenil 0.2mg, intravenous

Efficacy evaluation :

1. Determination of the impact of clobazam:

   * on the size of the area of secondary hyperalgesia induced by an UVB irradiation of the skin (sunburn model). The area is mapped with an electronical Von Frey filament
   * on the pain threshold (heat, static and mechanical threshold) in the primary and secondary area of hyperalgesia
   * on the nociceptive flexion reflex
   * on tolerance pain threshold (cold pressor test)
   * on the degree of sedation measured by saccadic eye movements, digit substation symbols test (DSST) and numerical rating scale.
2. Determination of the concentration-time curve of clobazam and PK-PD modelling.

Statistical Methods :

Based on the results of a previous study done in our unit, assessing the effect of the association of paracetamol and ketorolac on the sunburn model30, the number of volunteers required to detect a 30% reduction in the area of hyperalgesia is 4830. However we chose a lower intensity of UVB irradiation than in previous studies. Using a dose of irradiation of 3 med , this number falls to 18, adopting a 5% level for statistical significance and a 80% power. Taking these two results in account we will go for 25 volunteers.

Data will be analysed by multifactorial analysis of variance (MANOVA) and by analysis of variance (ANOVA) with repeated measures In the case of withdrawal, the data obtained will not be used in the analysis. Data set will however be completed by enrolling a substitute volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Male subject, age between 18 and 60 year old
* Caucasian
* Type 3 skin phototype
* Non smoker or moderate smoker (< 10 cigarettes/day)
* No clinically abnormal findings on history and/or on physical examination
* Presence of an area of secondary hyperalgesia after UVB irradiation

Exclusion Criteria:

* Any concomitant illness
* Current or past history of drug and alcohol abuse or current intake of more than 3 glasses of alcohol a day or more than 21 glasses of alcohol per week
* Psychotropic drug intake during the last month
* Sun allergy or any skin disease
* Current and regular intake of any drugs that might affect nociception Paracetamol, or NSAIDS with a short half lives are permitted but should be stopped at least 48 h before the UVB session

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Determination of the impact of clobazam on the change in the area of secondary hyperalgesia (in cm2) mapped with a Von Frey filament (256mN). | 3 single days spaced out with at least two weeks wash-out periods

SECONDARY OUTCOMES:
Change in the pain threshold (heat (°C) static mechanical (g) and dynamic mechanical (Numerical rating scale NAS) in the area of secondary hyperalgesia | 3 single days spaced out with at least two weeks wash-out periods
Change in the pain threshold (heat (°C ) static mechanical (g) and dynamic mechanical (NAS)) in the area of primary hyperalgesia | 3 single days spaced out with at least two weeks wash-out periods
Change in Nociceptive Flexion Reflex | 3 single days spaced out with at least two weeks wash-out periods
Change in the latency and in the area under the pain intensity/time curve in cold pressor test | 3 single days spaced out with at least two weeks wash-out periods
Change in mean target saccades peak velocity, target saccades acceleration and deceleration, in saccade latency (msec), in saccadic accuracy, in smooth pursuit lead time and in the number of saccadic intrusions in the smooth pursuit. | 3 single days spaced out with at least two weeks wash-out periods
Change in the total number and in the correct number of symbols drawn in the DDST challenge. | 3 single days spaced out with at least two weeks wash-out periods
Time concentration curve evaluation: blood samples at 0,5, 1, 2, 4, 6, 8,12, and at 24 hours post-dose | 3 single days spaced out with at least two weeks wash-out periods
  Clobazam and N-desmethylclobazam concentrations (µg/mL)
Pharmacokinetic/ pharmacodynamic modelling. | 3 single days spaced out with at least two weeks wash-out periods

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals, Geneva, Switzerland